CLINICAL TRIAL: NCT03801993
Title: Multicenter Study of Patient-reported Gastrointestinal Symptoms in People With Cystic Fibrosis (GALAXY-OB-18)
Brief Title: Multicenter Study of Patient-reported Gastrointestinal Symptoms in People With Cystic Fibrosis
Acronym: GALAXY
Status: Completed | Type: Observational
Sponsor: Chris Goss (Other)
Collaborators: Emory University (Other); University of North Carolina, Charlotte (Other); University of Texas (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Chris Goss, Professor of Medicine and Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: GALAXY-OB-18
Record Dates: First submitted 2019-01-04; First posted 2019-01-14 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; GI; nutrition; quality of life; bowel; constipation; gastrointestinal
MeSH Terms: conditions — Cystic Fibrosis; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Subjects: Subjects with a diagnosis of Cystic Fibrosis (CF) who meet all the inclusion and none of the exclusion criteria will be eligible for participation in this study.

SUMMARY:
This is a prospective, multicenter, observational study designed to collect gastrointestinal related data in patients with Cystic Fibrosis (CF).

DETAILED DESCRIPTION:
There are currently no large, multicenter prospective clinical trials examining management of constipation or other gastrointestinal (GI) symptoms in people with cystic fibrosis (CF). Current recommendations in the CF literature are largely based on expert consensus and opinions. Yet, constipation and other GI symptoms are crucial factors in quality of life (QOL) and maintenance of optimal nutritional state in people with CF. This study will use GI-symptomatology questionnaires to understand the multiple overlapping GI symptoms in people with CF.

Eligible subjects will be consented and enrolled in the study at the Enrollment Visit. At the visit, the subject or parent/guardian will complete the patient reported outcome surveys (PROs) using a mobile device (e.g., smartphone or tablet). The same questionnaires will be completed on a mobile device outside the clinic three additional times. The PROs will consist of four questionnaires: Patient Assessment of Constipation Symptoms (PAC-SYM), Patient Assessment of Gastrointestinal Symptoms (PAGI-SYM), Patient Assessment of Constipation Quality of Life (PAC-QOL) and a disease-specific questionnaire (Bristol Stool Scale and questions about fecal incontinence, and stool quality and frequency).

ELIGIBILITY:
Inclusion Criteria:

1. All genders ≥ 2 years of age at time of consent
2. Documentation of a Cystic Fibrosis (CF) diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   * Sweat chloride equal to or greater than 60 milliequivalent (mEq)/liter by quantitative pilocarpine iontophoresis test (QPIT)
   * Two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
   * Abnormal nasal potential difference (NPD) (change in NPD in response to a low chloride solution and isoproterenol of less than -5 mV)
3. Enrolled in the Cystic Fibrosis Foundation Patient Registry (subjects may enroll in the Registry at Enrollment Visit if not previously enrolled)
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative
5. Willing to complete questionnaires on mobile device
6. Able to use the Medidata Patient Cloud mobile application for completing the questionnaires

Exclusion Criteria:

1. Presence of a condition or abnormality that, in the opinion of the Investigator, would complicate interpretation of study outcome data or interfere with achieving the study objectives
2. Presence of a pulmonary exacerbation at the Enrollment Visit
3. Hospitalization for distal intestinal obstruction syndrome (DIOS) within the 28 days prior to the Enrollment Visit
4. Current gastrointestinal (GI) or abdominal/pelvic malignancy
5. Abdominal or pelvic surgery within the 28 days prior to the Enrollment Visit
6. At the time of the Enrollment Visit, planned abdominal or pelvic surgery or bowel cleanout in the 28 days after the Enrollment Visit
7. Initiation of new CFTR modulator therapy within the 4 weeks prior to the Enrollment Visit
8. Intent to initiate new CFTR modulator therapy within 28 days of the Enrollment Visit

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a diagnosis of Cystic Fibrosis (CF) who meet all the inclusion and none of the exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Jay Freeman, MD, MSc, Principal Investigator — Emory University/Children's Healthcare; Baharak Moshiree, MD, Principal Investigator — University of North Carolina Charlotte, Atrium Health; Meghana Sathe, MD, Principal Investigator — University of Texas Southwestern/Children's Health
Locations (26):
- United States (26):
  - Stanford University Medical Center, Palo Alto, California
  - Central Connecticut Cystic Fibrosis Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta and Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Atrium Health Pulmonary Care, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma Cystic Fibrosis Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - Intermountain Cystic Fibrosis Center, Salt Lake City, Utah
  - The Children's Specialty Center Fletcher Allen Health Care, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moshiree B, Freeman AJ, Vu PT, Khan U, Ufret-Vincenty C, Heltshe SL, Goss CH, Schwarzenberg SJ, Freedman SD, Borowitz D, Sathe M; GALAXY Study Group. Multicenter prospective study showing a high gastrointestinal symptom burden in cystic fibrosis. J Cyst Fibros. 2023 Mar;22(2):266-274. doi: 10.1016/j.jcf.2022.10.006. Epub 2022 Oct 29. PMID 36319569

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled: Eligible participant who fully completed at least one ePRO at Baseline Visit
Period: Overall Study
Arm/Group | All Enrolled
Started (With 400 subjects, this study will allow estimation of variability (between and within subject) in 160 pediatric subjects and 240 adult subjects.) | 402
Week 1 (At least one fully completed ePRO at Week 1) | 329
Week 2 (At least one fully completed ePRO at Week 2) | 324
Week 4 (At least one fully completed ePRO at Week 4) | 312
Completed (Fully completed at least one ePRO at all Follow-up Weeks) | 254
Not Completed | 148

BASELINE CHARACTERISTICS:
Groups:
- Age <18: Age <18 years at baseline among All Enrolled
- Age >=18: Age >= 18 years at baseline among All Enrolled
- Total: Total of all reporting groups
Arm/Group | Age <18 | Age >=18 | Total
Number analyzed (Participants) | 169 | 233 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 169 | 0 | 169
  Between 18 and 65 years | 0 | 233 | 233
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 10.28 [2.09 to 17.83] | 26.23 [18.04 to 61.13] | 19.36 [2.09 to 61.13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 118 | 193
  Male | 94 | 115 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 157 | 226 | 383
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 164 | 218 | 382
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 3 | 4
Genotype [Count of Participants; unit: Participants] — Genotype was extracted by medical record review reporting prior results of tests for the diagnosis of cystic fibrosis. The variant F508del is common, and participants having one copies (F508del Heterozygous), no copies (Other), or without genetic test results (Unknown) have more heterogeneous phenotypes than those with two copies (F508del Homozygous).
  Participants
    F508 Heterozygous | 64 | 78 | 142
    F508 Homozygous | 89 | 126 | 215
    Other/Unknown | 16 | 29 | 45
Mutation Class [Count of Participants; unit: Participants] — Each of a patient's allele genotype variants were matched to traditional CFTR mutation classifications: Protein production (Class I), Protein processing (Class II), Gating (Class III), Conduction (Class IV), and Insufficient protein (Class V). The maximum class was assigned to the genotype pair and grouped by severity, with Class I-III "more severe" and Class IV-V "less severe". Unmatched variants were assigned class Unknown. F508del for example is Class II, so a participant heterozygous for F508del would have mutation Class II or greater, depending on the other allele variant's class.
  Participants
    I-III (more severe) | 129 | 185 | 314
    IV-V (less severe) | 13 | 17 | 30
    Unknown | 27 | 31 | 58
Sweat Chloride at Diagnosis [Mean (Standard Deviation); unit: mEq/L] | 91.00 (22.08) | 97.53 (18.05) | 94.73 (20.11)
Pancreatic Sufficiency [Count of Participants; unit: Participants]
  Insufficient | 149 | 204 | 353
  Sufficient | 20 | 29 | 49
Modulator Use [Count of Participants; unit: Participants]
  None | 87 | 87 | 174
  Ivacaftor | 10 | 10 | 20
  Lumacaftor/Ivacaftor | 55 | 38 | 93
  Tezacaftor/Ivacaftor | 16 | 87 | 103
  Triple Combination | 1 | 10 | 11
  Ivacaftor and Triple Combination | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Fully Completed at Least One ePRO
Description: Number participants with scheduled outside-the-clinic assessments who fully completed at least one of the four PROs. A "fully complete" questionnaire is defined as having responded to all questions with no missing responses.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Age <18 | Age >=18
Number analyzed (Participants) | 169 | 233
Participants
  Week 1 | 133 | 196
  Week 2 | 130 | 194
  Week 4 | 125 | 187

2. Secondary Outcome: Number of Participants With Period-Prevalence of Constipation
Description: This table summarizes the period-prevalence of protocol-defined constipation. For each follow-up response, constipation was defined by the protocol as having fewer than 3 bowel movements and/or Bristol Stool Scale of Type 1 or 2 (hard lumps) in the past 7 days. Period prevalence is defined as occurrence of the symptom at any time from baseline to week 4. Only participants who fully completed the disease-specific questionnaire at baseline and all follow-up weeks were considered.
Time Frame: 1 month
Population: Participants who fully completed the disease-specific questionnaire at baseline and all follow-up weeks
Measure: Count of Participants; unit: Participants
Groups:
- Age <18 With Complete Follow-up: Participants under 18 years old at baseline who fully completed the disease-specific questionnaire at baseline and all follow-up weeks were considered.
- Age >=18 With Complete Follow-up: Participants 18 years or older at baseline who fully completed the disease-specific questionnaire at baseline and all follow-up weeks were considered.
Arm/Group | Age <18 With Complete Follow-up | Age >=18 With Complete Follow-up
Number analyzed (Participants) | 95 | 151
Participants | 18 | 35

3. Secondary Outcome: Mean Patient Reported Outcome (PRO) Scores
Description: Mean PRO scores (PAC-SYM score range: 0-4, PAGI-SYM score range: 0-5, PAC-QOL score range: 0-4) at time of enrollment (Visit 1) where lower scores correspond to less symptom severity.
Time Frame: At Visit 1 (1 day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Age <18 | Age >=18
Number analyzed (Participants) | 169 | 233
score on a scale
  PAC-SYM Total Score | 0.49 (0.45) | 0.64 (0.55)
  PAGI-SYM Total Score | 0.49 (0.56) | 0.78 (0.66)
  PAC-QOL Total Score | 0.58 (0.47) | 0.73 (0.59)

4. Secondary Outcome: Number of Participants Treated for GI Symptoms
Description: Number of enrolled participants receiving treatment for GI symptoms at Visit 1
Time Frame: At Visit 1 (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Age <18 | Age >=18
Number analyzed (Participants) | 169 | 233
Participants
  Initiating or Receiving GI Treatment | 167 | 228
  GI Treatment for Constipation | 88 | 78
  GI Treatment for Non-Constipation | 166 | 228
  Use GI Tube | 24 | 8
  On Azithromycin | 60 | 131
  On drugs used in diabetes | 12 | 59

ADVERSE EVENTS:
Time Frame: Adverse Events, including Deaths and Serious Adverse Experiences, were not collected or monitored as part of this study.
Description: Adverse Events, including Deaths and Serious Adverse Experiences, were not collected or monitored as part of this study.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03801993/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03801993/SAP_001.pdf